CLINICAL TRIAL: NCT04193839
Title: Reducing Errors In The Neonatal Intensive Care Unit. The SAPHET-i Study: Secure, Automated, Functional, High-Tech Therapeutic Approach for iNFANTS
Brief Title: Reducing Errors In The Neonatal Intensive Care Unit
Acronym: SAPHET-i
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Poliambulanza Istituto Ospedaliero (Other)
Responsible Party: Principal Investigator, Maria Pierro, Principal investigator, Fondazione Poliambulanza Istituto Ospedaliero
Other Study IDs: NP 3751
Record Dates: First submitted 2019-11-28; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Medication Errors and Other Product Use Errors and Issues; Adverse Drug Event
Keywords: Computerized Provider Order entry; Patient safety; Quality improvement; Medication errors; Adverse events; Bar code medication administration; Neonates
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Medical Order Entry Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paper Order Entry cohort: Patients admitted to the NICU during the pre-intervention phase, enrolled in the study after parental consent. The medications prescribed to the patients enrolled during the pre-intervention period will be handled with the paper order entry
- CPOE + BCMA cohort: Patients admitted to the NICU during the post-intervention phase, enrolled in the study after parental consent. The medications prescribed to the patients enrolled during the post-intervention period will be handled with the Computerized Provider Order Entry + Bar Code Medication Administration (BCMA)
  Interventions: Other: Computerized Provider Order Entry (CPOE) plus Bar Code Medication Administration (BCMA)

INTERVENTIONS:
Other: Computerized Provider Order Entry (CPOE) plus Bar Code Medication Administration (BCMA) — Computerized provider order entry (CPOE) refers to the process of providers entering and sending treatment instructions - including medication, laboratory, and radiology orders - via a computer application rather than paper, fax, or telephone. The bar Code Medication Administration (BCMA) is a system that consists of a bar code reader, a portable or desktop computer with wireless connection, a computer server, and some software. Before the administration of medications to the patients the patient unique barcode identification is scanned in order to verify the patient's identity.
  Groups: CPOE + BCMA cohort

SUMMARY:
This is a monocentric prospective pre and post-intervention study, aiming at analyzing the efficacy of the Computerized Provider Order Entry (CPOE) plus Bar Code Medication Administration (BCMA) as compared to paper order entry in reducing medication erros (MEs) in the Neonatal Intensive Care Unit (NICU)

DETAILED DESCRIPTION:
Medication errors are a burden to the health care system. The neonatal population, in particular the infants admitted to the NICU, are at higher risk of MEs as compared to the adult and pediatric population. Moreover adverse events (ADEs) occur more frequently and may be particularly severe in neonates.

Several strategies have been tried in order to decrease the incidence of MEs in the NICU. Among these, some studies investigated the effectiveness of CPOE in reducing MEs in hospitalised patients. However, results have been inconsistent. So far, no study investigated the association of CPOE + BCMA in neonates.

The investigators designed a monocentric prospective pre and post-intervention observational study to investigate the efficacy of the CPOE plus BCMA as compared to paper order entry in reducing MEs in the NICU population.

ELIGIBILITY:
Inclusion criteria:

* Admission to the NICU
* Need of pharmacological intervention
* Informed parental consent

Exclusion criteria:

* Lack of parental consent

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any patient admitted to the NICU who needs pharmacological intervention is eligible.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of medication errors | From date of NICU admission up to discharge, up to 18 months
  The investigators will record all types of errors (prescription, transcription, preparation, administration errors) through spontaneous reporting, structured daily audit and chart revision

SECONDARY OUTCOMES:
Number of preventable adverse drug events | From date of NICU admission up to discharge, up to 18 months
  The investigators will record the number of preventable and non preventable adverse drug events

CONTACTS AND LOCATIONS:
Overall Officials: Maria Pierro, MD, PhD, Principal Investigator — Fondazione Poliambulanza Istituto Ospedaliero
Locations (1):
- Fondazione Poliambulanza Istituto Ospedaliero, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Undecided